CLINICAL TRIAL: NCT00450450
Title: A Phase III Randomized Trial of G-CSF Stimulated Bone Marrow vs. Conventional Bone Marrow as a Stem Cell Source In Matched Sibling Donor Transplantation
Brief Title: Donor Bone Marrow Transplant With or Without G-CSF in Treating Young Patients With Hematologic Cancer or Other Diseases
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASCT0631; NCI-2009-01069 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ASCT0631 (Other: Children's Oncology Group); COG-PBMTC-STC051 (Other: Children's Oncology Group); CDR0000532926 (Other: Clinical Trials.gov); U10CA098543 (NIH)
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Results first posted 2017-05-09 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2021-06

CONDITIONS: Childhood Acute Lymphoblastic Leukemia in Remission; Childhood Acute Myeloid Leukemia in Remission; Childhood Chronic Myelogenous Leukemia; Childhood Myelodysplastic Syndromes; Chronic Phase Chronic Myelogenous Leukemia; de Novo Myelodysplastic Syndromes; Juvenile Myelomonocytic Leukemia; Previously Treated Myelodysplastic Syndromes; Recurrent Childhood Acute Lymphoblastic Leukemia; Secondary Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelomonocytic, Juvenile; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Transplantation; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients undergo filgrastim (G-CSF)-stimulated allogeneic bone marrow transplantation on day 0.
  Interventions: Procedure: allogeneic bone marrow transplantation; Other: laboratory biomarker analysis; Biological: filgrastim
- Arm II (Active Comparator): Patients undergo conventional allogeneic bone marrow transplantation on day 0.
  Interventions: Procedure: allogeneic bone marrow transplantation; Other: laboratory biomarker analysis

INTERVENTIONS:
Procedure: allogeneic bone marrow transplantation — Patients undergo allogeneic BMT
  Other Names: bone marrow therapy, allogeneic; bone marrow therapy, allogenic; transplantation, allogeneic bone marrow; transplantation, allogenic bone marrow
Other: laboratory biomarker analysis — Correlative studies
Biological: filgrastim — Given IV
  Other Names: Granulocyte Colony-Stimulating Factor; r-metHuG-CSF; G-CSF; Neupogen; NSC #614629
  Arms: Arm I

SUMMARY:
This randomized phase III trial is studying donor bone marrow transplant with or without G-CSF to compare how well they work in treating young patients with hematologic cancer or other diseases. Giving chemotherapy and total-body irradiation before a donor bone marrow transplant helps stop the growth of cancer or abnormal cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving methotrexate and tacrolimus or cyclosporine before and after transplant may stop this from happening. It is not yet known whether donor bone marrow transplant is more effective with or without G-CSF in treating hematologic cancer or other diseases.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Compare improvement in event-free survival of patients with hematologic cancer or other diseases undergoing filgrastim (G-CSF)-stimulated bone marrow transplantation (BMT) vs conventional BMT.

SECONDARY OBJECTIVES:

I. Compare the incidence and time to engraftment in patients treated with these regimens.

II. Compare rates of acute and chronic graft-vs-host disease (GVHD) in patients treated with these regimens.

III. Correlate incidence of acute and chronic GVHD with absolute T-cell numbers, Th1 vs Th2 profile of T cells, dendritic cell populations, and T-regulatory cell content.

IV. Assess the impact of G-CSF-stimulated BMT as a stem cell source on hospital stay and treatment-related mortality at day 100 in patients treated with this regimen.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to risk (high vs intermediate vs standard).

CONDITIONING REGIMEN: Co-enrolled on COG-ASCT0431 or COG-AAML0531; Patients receive a conditioning regimen as defined on that treatment study.

ACUTE LYMPHOBLASTIC LEUKEMIA (ALL): Patients undergo total-body irradiation (TBI) twice daily on days -8 to -6. Patients receive thiotepa IV on days -5 and -4 and high-dose cyclophosphamide IV over 1 hour on days -3 and -2. Some patients with CNS leukemia or very high-risk ALL in first complete remission receive cranial radiotherapy.

ACUTE MYELOID LEUKEMIA, JUVENILE MYELOMONOCYTIC, CHRONIC MYELOGENOUS LEUKEMIA, OR MYELODYSPLASTIC SYNDROMES: (myeloid malignancies) Patients receive busulfan IV over 2 hours every 6 hours on days -9 to -6 and high-dose cyclophosphamide IV over 1 hour on days -5 to -2.

GRAFT-VS-HOST DISEASE (GVHD) PROPHYLAXIS: Co-enrolled on COG-ASCT0431 or COG-AAML0531: Patients undergo GVHD prophylaxis as defined on that treatment study.

ALL: Patients receive tacrolimus IV or orally beginning on day -2 and continuing until day 42, followed by a taper until day 98. Patients also receive methotrexate IV on days 1, 3, and 6.

MYELOID MALIGNANCIES: Patients receive cyclosporine IV continuously or orally beginning on day -1 and continuing until day 42 or day 50, followed by a taper for 8-16 weeks. Patients also receive methotrexate IV on days 1, 3, 6, and 11.

ALLOGENEIC BONE MARROW TRANSPLANTATION (BMT): Patients are randomized to 1 of 2 transplantation arms.

ARM I: Patients undergo filgrastim (G-CSF) -stimulated allogeneic BMT on day 0.

ARM II: Patients undergo conventional allogeneic BMT on day 0.

After completion of study treatment, patients are followed at 1 year and then annually for 5-10 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hematologic cancer or other disease, including any of the following:

  * Chronic myelogenous leukemia in first or second chronic phase
  * Acute lymphoblastic leukemia (ALL), meeting any of the following criteria:

    * Relapsed ALL enrolled on a Children's Oncology Group (COG) relapse clinical trial OR received ≥ 1 round of reinduction therapy (4-6 weeks) and 1 round of intensive consolidation chemotherapy (3-6 weeks)
    * ALL in second complete remission (CR)* after a bone marrow, extramedullary, or combined bone marrow and extramedullary relapse
    * Very high-risk ALL in first CR, defined as any of the following:

      * Philadelphia chromosome-positive ALL
      * Hypodiploidy (< 44 chromosomes)
      * Mixed lineage leukemia rearrangement
      * Induction failure
  * Acute myeloid leukemia in first or second CR

    * Induction therapy must be completed
  * Juvenile myelomonocytic leukemia
  * Myelodysplastic syndromes
* No clinically evident CNS or extramedullary disease
* No blasts seen on cerebrospinal fluid cytospin
* Post-relapse reinduction therapy must be completed
* Not planning to receive reduced-intensity conditioning regimen
* Not planning to receive a graft that has undergone T-cell depletion
* No Down syndrome
* Matched sibling donor must be available and must be enrolled on ASCT0631D companion study
* Karnofsky performance status (PS) 60-100% (patients > 16 years of age) OR Lansky PS 60-100% (patients ≤ 16 years of age)
* AST or ALT < 5 times upper limit of normal for age
* Bilirubin < 2.5 mg/dL (unless due to Gilbert's syndrome)
* Creatinine clearance or radioisotope glomerular filtration rate ≥ 70 mL/min OR serum creatinine base on age and/or gender as follows:

  * 0.4 mg/dL (1 month to < 6 months of age)
  * 0.5 mg/dL (6 months to < 1 year of age)
  * 0.6 mg/dL (1 to 2 years of age)
  * 0.8 mg/dL (2 to < 6 years of age)
  * 1.0 mg/dL (6 to < 10 years of age)
  * 1.2 mg/dL (10 to < 13 years of age)
  * 1.5 mg/dL (male) or 1.4 mg/dL (female) (13 to < 16 years of age)
  * 1.7 mg/dL (male) or 1.4 mg/dL (female) (≥ 16 years of age)
* Shortening fraction ≥ 27% by echocardiogram OR LVEF ≥ 50% by radionuclide angiogram
* FEV_1, FVC, and DLCO ≥ 60% OR meets the following criteria (for patients unable to cooperate for pulmonary function tests):

  * No evidence of dyspnea at rest
  * No exercise intolerance
  * No requirement for supplemental oxygen therapy
* Not pregnant or nursing
* No known HIV
* No known uncontrolled fungal, bacterial, or viral infections

  * Patients acquiring fungal disease during induction therapy may proceed if they have a significant response to antifungal therapy with no or minimal evidence of disease remaining by CT scan
* No prior allogeneic or autologous stem cell transplantation

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2007-12-31 (Actual); Primary Completion 2013-06-01 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan A. Grupp, MD PhD, Principal Investigator — Children's Oncology Group
Locations (21):
- United States (21):
  - Children's Oncology Group, Arcadia, California
  - University of California San Francisco Medical Center-Parnassus, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Childrens Memorial Hospital, Chicago, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - Kosair Children's Hospital, Louisville, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York Medical College, Valhalla, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Control BM Arm: Conventional bone marrow transplant (BM)
- Experimental G-BM Arm: G-CSF (filgrastim) stimulated bone marrow (G-BM)
Period: Overall Study
Arm/Group | Control BM Arm | Experimental G-BM Arm
Started | 13 | 14
Completed | 8 | 11
Not Completed | 5 | 3
Not completed — Death | 1 | 3
Not completed — Relapse | 2 | 0
Not completed — Missing Data | 2 | 0

BASELINE CHARACTERISTICS:
Population: Group 2 enrollment total is 14, patient 774353 enrolled on study, but was not randomized and didn't contribute any data. Group 2 AE total is 13.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control BM Arm | Experimental G-BM Arm | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Continuous [Median (Full Range); unit: Whole year] | 12 [0 to 20] | 11 [3 to 20] | 12 [0 to 20]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 8 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 11 | 11 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: Participants]
  United States | 12 | 14 | 26
  Australia | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Estimated Two-year Event-free Survival (EFS)
Description: EFS is defined as relapse or treatment-related mortality (TRM). relapse is defined by either morphological or cytogenetic evidence of ALL consistent with pre-transplant features.
Time Frame: at 2 years
Population: Early terminated study. One patient is inevaluable for EFS on experimental arm and is excluded from analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Control BM Arm | Experimental G-BM Arm
Number analyzed (Participants) | 13 | 13
Percentage of patients | 66 [32 to 86] | 83 [47 to 96]

2. Secondary Outcome: Estimated Graft Failure Rate
Description: Primary graft failure is defined as the failure to achieve an absolute neutrophil count of more than 5000 per cubic millimeter for at least three consecutive days by Day +42.
Time Frame: Up to 10 years
Population: One patient is inevaluable for EFS on experimental arm and is excluded from analysis.
Measure: Number; unit: Percentage of patients
Arm/Group | Control BM Arm | Experimental G-BM Arm
Number analyzed (Participants) | 13 | 13
Percentage of patients | 0 | 0

3. Secondary Outcome: Estimated Incidence of Grade III-IV Acute Graft-versus-host Disease (aGVHD)
Description: Stage III-IV aGVHD is defined as: Stage 0-3 skin, with Stage 2-3 liver, or Stage 2-3 GI; OR Stage 4 skin, liver or GI involvement.
Time Frame: Up to 3 months
Population: One patient is inevaluable and is excluded from analysis.
Measure: Number; unit: Percentage of patients
Arm/Group | Control BM Arm | Experimental G-BM Arm
Number analyzed (Participants) | 13 | 13
Percentage of patients | 7.69 | 15.38

4. Secondary Outcome: Estimated 100-day Transplant Related Mortality (TRM) Percentage
Description: Death in a patient after transplant due to protocol treatment is defined as an TRM.
Time Frame: 100 days
Population: One patient is inevaluable and is excluded from analysis.
Measure: Number; unit: percentage of patients
Arm/Group | Control BM Arm | Experimental G-BM Arm
Number analyzed (Participants) | 13 | 13
percentage of patients | 0 | 7.69

5. Secondary Outcome: Estimated Percentage of Chronic Graft-versus-host Disease (cGVHD)
Description: cGVHD definition is based on BMT CTN MOP SEPT. 2005; outlined in Protocol Appendix III.
Time Frame: 18 months post-transplant
Population: Included only patients survived beyond 100 days.
Measure: Number; unit: percentage of patients
Arm/Group | Control BM Arm | Experimental G-BM Arm
Number analyzed (Participants) | 13 | 12
percentage of patients | 7.69 | 0

6. Secondary Outcome: Estimated Median Time to Neutrophil Engraftment
Description: Median Time from transplant to neutrophil engraftment
Time Frame: Up to 10 years
Population: One patient was inevaluable and excluded from the analysis.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Control BM Arm | Experimental G-BM Arm
Number analyzed (Participants) | 13 | 13
Days | 23 [20 to 25] | 20 [16 to 23]

7. Secondary Outcome: Estimated Median Length of Initial Hospitalization
Description: Estimated and compared between randomization arms using the Wilcoxon rank-sum test.
Time Frame: Up to 10 years
Population: Data regarding length of Initial Hospitalization are not collected for this study according to Study Chair.
Arm/Group | Control BM Arm | Experimental G-BM Arm
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Immune Reconstitution
Description: Summarized graphically. Generalized estimating equation will be used to model the levels as a function of time and randomization assignment and to test the impact of G-CSF stimulation on immune reconstruction.
Time Frame: Up to 1 year
Population: Data are not collected for this study.
Arm/Group | Control BM Arm | Experimental G-BM Arm
Number analyzed (Participants) | 0 | 0

9. Other Pre Specified Outcome: Infused Nucleated and CD34+ Cell Doses
Description: Compared using the Wilcoxon rank-sum test.
Time Frame: Up to 10 years
Population: Data are not collected for this study.
Arm/Group | Control BM Arm | Experimental G-BM Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Group 2 enrollment total is 14, patient 774353 enrolled on study, but was not randomized and didn't contribute any data. Group 2 AE total is 13.
Arm/Group | Control BM Arm | Experimental G-BM Arm
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/13
Other Adverse Events (participants affected / at risk) | 8/13 | 7/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control BM Arm (N=13) | Experimental G-BM Arm (N=13)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control BM Arm (N=13) | Experimental G-BM Arm (N=13)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 4 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 2
Autoimmune disorder (Immune system disorders) | 0 | 1
Bladder infection (Infections and infestations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 1
Death NOS (General disorders) | 0 | 1
Edema face (General disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 2 | 0
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 2
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 5 | 0
Lung infection (Infections and infestations) | 1 | 0
Lymphocyte count decreased (Investigations) | 2 | 1
Mucositis oral (Gastrointestinal disorders) | 2 | 3
Multi-organ failure (General disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 5 | 3
Oral pain (Gastrointestinal disorders) | 1 | 1
Peripheral nerve infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Platelet count decreased (Investigations) | 5 | 5
Rectal mucositis (Gastrointestinal disorders) | 0 | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
White blood cell decreased (Investigations) | 5 | 2

LIMITATIONS AND CAVEATS:
ASCT0631 is closed to further patient entry as of 11/25/2011 due to poor accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.